CLINICAL TRIAL: NCT06510712
Title: Nutritional Risk and Health Research for Hospitalized Patients With Neurology Disorders in China
Brief Title: Nutritional Risk for Hospitalized Patients With Neurology Disorders in China
Status: Not yet recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: X-MEC-2024-001
Record Dates: First submitted 2024-07-14; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Neurological Disorder
Keywords: nutrition; the risk of malnutrition
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neurology disorders are one of the major public health problems that seriously threaten human health. It often accompanied by various nutritional problems, which can aggravate the primary disease, lead to serious complications, prolong the hospitalization, lead to poor prognosis, and increase family and social economic burdens. According to the previous studies, the risk of malnutrition was approximately 58.5% of stroke patients, and 6% had moderate to severe malnutrition in China. Another study conducted in Beijing showed that the risk of malnutrition of elderly patients in the department of neurology was significantly higher than in other departments (28.5% vs. 26.4%). Strengthening nutritional supervision of patients with neurology disorders will benefit to improve patients' prognosis. Therefore, the aim of this study is to investigate the nutritional status of inpatients with neurology disorders in China, evaluate the impact of different nutritional status on patients' health outcomes, and establish a high-quality, standardized nutrition and health cohort database for neurology disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. The primary diagnosis was neurological disorders;
3. Written informed consent.

Exclusion Criteria:

1. Life expectancy is < 3 months;
2. Researchers think other ineligible participant for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with the primary diagnosis are neurological disoders
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 30 days
  Mortality defined as all-cause mortality from inclusion to day 30

SECONDARY OUTCOMES:
ICU admission | 30 days
  ICU admission defined as admission to the intensive care unit from the medical ward from inclusion to day 30
Non-elective hospital readmission | 30 days
  Non-elective hospital readmission defined as non-scheduled hospital readmission after discharge from the index hospital stay to day 30
Major complications | 30 days
  Major complications defined as the following complications occurring from inclusion (i.e., not present at the time of inclusion) to day 30 I. Adjudicated nosocomial infection or abscess requiring antibiotic treatment II. respiratory failure with need for invasive or non-invasive ventilation III. major cardiovascular events including stroke, intracranial bleeding, cardiac arrest, myocardial infarction with and without invasive procedure and pulmonary embolism IV. acute renal failure (defined by 2x increase of baseline creatinine or new requirement of dialysis do to volume overload or electrolyte disturbance) V. gastro-intestinal events (hemorrhage, intestinal perforation)
Decline in functional status of 10% or more | 30 days
  decline in functional status of 10% or more from admission to day 30 measured by the Barthel's index.
length of in hospital days | 30 days
  Total length of in hospital days 30 days

OTHER OUTCOMES:
Adverse events | 30 days
  Each of the adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Junwei Hao, PhD, Principal Investigator — Capital Medical University Xuanwu Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] GBD 2019 Stroke Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Neurol. 2021 Oct;20(10):795-820. doi: 10.1016/S1474-4422(21)00252-0. Epub 2021 Sep 3. PMID 34487721
- [Background] Wang YJ, Li ZX, Gu HQ, Zhai Y, Jiang Y, Zhao XQ, Wang YL, Yang X, Wang CJ, Meng X, Li H, Liu LP, Jing J, Wu J, Xu AD, Dong Q, Wang D, Zhao JZ; China Stroke Statistics 2019 Writing Committee. China Stroke Statistics 2019: A Report From the National Center for Healthcare Quality Management in Neurological Diseases, China National Clinical Research Center for Neurological Diseases, the Chinese Stroke Association, National Center for Chronic and Non-communicable Disease Control and Prevention, Chinese Center for Disease Control and Prevention and Institute for Global Neuroscience and Stroke Collaborations. Stroke Vasc Neurol. 2020 Sep;5(3):211-239. doi: 10.1136/svn-2020-000457. Epub 2020 Aug 21. PMID 32826385
- [Background] Brenton JN, Lehner-Gulotta D, Woolbright E, Banwell B, Bergqvist AGC, Chen S, Coleman R, Conaway M, Goldman MD. Phase II study of ketogenic diets in relapsing multiple sclerosis: safety, tolerability and potential clinical benefits. J Neurol Neurosurg Psychiatry. 2022 Jun;93(6):637-644. doi: 10.1136/jnnp-2022-329074. Epub 2022 Apr 13. PMID 35418509
- [Background] FOOD Trial Collaboration. Poor nutritional status on admission predicts poor outcomes after stroke: observational data from the FOOD trial. Stroke. 2003 Jun;34(6):1450-6. doi: 10.1161/01.STR.0000074037.49197.8C. Epub 2003 May 15. PMID 12750536
- [Background] Mehta A, De Paola L, Pana TA, Carter B, Soiza RL, Kafri MW, Potter JF, Mamas MA, Myint PK. The relationship between nutritional status at the time of stroke on adverse outcomes: a systematic review and meta-analysis of prospective cohort studies. Nutr Rev. 2022 Nov 7;80(12):2275-2287. doi: 10.1093/nutrit/nuac034. PMID 35640017
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34487721/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32826385/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35418509/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/12750536/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35640017/